CLINICAL TRIAL: NCT02423863
Title: In Situ, Autologous Therapeutic Vaccination Against Solid Cancers With Intratumoral Hiltonol® (Poly-ICLC): An Adaptive, Multicenter, Phase II Clinical Study
Brief Title: In Situ, Autologous Therapeutic Vaccination Against Solid Cancers With Intratumoral Hiltonol®
Acronym: Poly-ICLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oncovir, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); Icahn School of Medicine at Mount Sinai (Other); Bay Hematology Oncology (Unknown); National Cancer Institute (NCI) (NIH); University of Missouri-Columbia (Other); Chevy Chase Regional Cancer Care Associates LLC (Unknown); Dermatologic Surgery Center of Washington LLC and Skin Cancer Treatment Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC2014-001; 1R44CA183075-01A1 (NIH)
Record Dates: First submitted 2015-04-13; First posted 2015-04-22 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2017-09

CONDITIONS: Melanoma; Head and Neck Cancer; Sarcoma; Non-Melanoma Skin Cancers
Keywords: Cancer; Immunotherapy; Intratumoral Injection; Multicenter Study; Autovaccination; Solid Tumors; anti-PD1; anti-PDL1
MeSH Terms: conditions — Melanoma; Head and Neck Neoplasms; Sarcoma; Neoplasms | interventions — poly ICLC; Nivolumab; pembrolizumab; atezolizumab; cemiplimab; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hiltonol Poly-ICLC (Experimental): Open labeled, non randomized adaptive 2-stage design protocol. 21 study subjects were enrolled in stage I of the protocol. Up to an additional 60 patients. . Enrolled study subjects will receive Poly-ICLC (Hiltonol®) treatment alone or in combination with anti-PD-1 (Nivolumab, Pembrolizumab or Cemiplimab) or anti-PD-L1 (Atezolizumab or Durvalumab) over 6 months as defined in study treatment described below. MRI or CT imaging will be done per SOC at screening, 3 and 6-month time points.
  For purposes of analysis patients enrolled in Stage II of this study will be prospectively identified at initial screening as belonging to statistical Cohorts A, B, or C, which are based on patient status with regard to aPD1/aPDL1 therapy at study entry, (PD, SD, or treatment naïve). For purposes of this study, patient status is considered to be the primary eligibility variable, although sub analyses will also consider histology and particular checkpoint blocker used when possible.
  Interventions: Biological: Hiltonol

INTERVENTIONS:
Biological: Hiltonol — Wk 1 Days 1, 3 and 5: Poly-ICLC (Hiltonol®) 1 mg (0. 5 ml) IntraTumoral (priming treatment course). Weeks 2-25 Poly-ICLC (Hiltonol®) 1 mg (0.5 ml) IM twice a week with a 48-72 hour interval between the two injections, AND either:
  No additional immunotherapy OR
  ONLY ONE of the Anti-PD1 or anti-PDL-1 regimens will be administered, per manufacturer's dosing and clinical oncologist's discretion as follows: (Not to be Administered on the same day as Poly-ICLC [Hiltonol®]) Either Nivolumab, OR Pembrolizumab, OR Atezolizumab, OR Cemiplimab, OR Durvalumab
  Other Names: Poly-ICLC; Nivolumab; Pembrolizumab; Atezolizumab; Cemiplimab; Durvalumab

SUMMARY:
The purpose of this study is to evaluate the safety of sequential intratumoral (IT) plus intramuscular (IM) Polyinosinic-polycytidylic acid stabilized with polylysine and carboxymethylcellulose (poly-ICLC, Hiltonol®) for treatment of study subjects with accessible solid tumors, with or without checkpoint blockers. Enrolled study subjects will receive Poly-ICLC (Hiltonol®) treatment alone or in combination with anti-PD-1 (Nivolumab, Pembrolizumab or Cemiplimab) or anti-PD-L1 (Atezolizumab or Durvalumab) over 6 months as defined in study treatment described below. MRI or CT imaging will be done per SOC at screening, 3 and 6-month time points.

DETAILED DESCRIPTION:
For purposes of analysis patients enrolled in Stage II of this study will be prospectively identified at initial screening as belonging to statistical Cohorts A, B, or C, which are based on patient status with regard to aPD1/aPDL1 therapy at study entry, (PD, SD, or treatment naïve) per section 11.5. For purposes of this study, patient status is considered to be the primary eligibility variable, although sub analyses will also consider histology and particular checkpoint blocker used when possible. Please see section 12 (Statistical Analysis) for further discussion.

Week 1 Days 1, 3 and 5: Poly-ICLC (Hiltonol®) 1 mg (0. 5 ml) IntraTumoral (priming treatment course).

Weeks 2-25:

1. Poly-ICLC (Hiltonol®) 1 mg (0.5 ml) IM twice a week with a 48-72 hour interval between the two injections, AND either:
2. No additional immunotherapy OR
3. ONLY ONE of the following Anti-PD1 or anti-PDL-1 regimens will be administered, per manufacturer's dosing and clinical oncologist's discretion as follows: (Not to be Administered on the same day as Poly-ICLC [Hiltonol®])

   * Either Nivolumab (Opdivo), OR
   * Pembrolizumab (Keytruda), OR
   * Atezolizumab (Tecentriq) OR
   * Cemiplimab (Libtayo) OR
   * Durvalumab (Imfinzi)

NOTE: It is recognized that some patients will have already been on anti-PD-1 or anti-PD-L1 at the time of study entry. Such patients will not have their checkpoint blocker therapy interrupted, but will be started on Poly-ICLC on week one, as above

If well tolerated they continue at full dose of 1 mg IM twice weekly through week 25. Anti-PD-1 or anti-PD-L1 per manufacturers package insert begins on week two and continues through week 25 or beyond per standard of care at physician's discretion. After the end of Poly-ICLC treatment at week 25, aPD1 or aPDL1 can be continued at the discretion of the patient and treating physician, per SOC, independent of this protocol.

At week 26 study subjects will be assessed and response determined using the RECIST 1.1 criteria. This will include measurement of accessible lesions as well as CT scan of the chest, abdomen and pelvis and extremities or neck to assess for response, using RECIST 1.1. MRI of the brain may also be obtained as part of clinical follow of their disease, if clinically indicated as per standard clinical protocol. Study subject's response will be defined as BOR (CR, PR, SD) or PD. If tumors are present and accessible, biopsies of the injected tumor as well as of a non-targeted/non-injected tumor will also be obtained at week 26.

Study subjects with CR, PR, or SD may be offered an additional treatment cycle depending on study subject's health status, costs and/or drug availability. At week 26 a repeat tumor assessment will be performed, an optional biopsy may be performed.

Follow up Period:

After completion of study treatment, study subjects may be contacted by telephone at least twice over 12 months, or longer with patient consent to inquire on their health status (e.g., alive, remission, progressive disease, on new cancer treatment). Study subjects with an initial tumor response but then long-term recurrence during the follow up period may be offered additional cycles of treatment depending on the study subject's health status, costs and/or drug availability.

ELIGIBILITY:
Inclusion Criteria:

1)1) Histologically confirmed diagnosis of one of the following:

1. Melanoma
2. Squamous head and neck cancer
3. Sarcoma
4. Non-Melanoma skin cancers 2) Sarcoma Patients must be 14 years of age or older. All other patients must be 18 years of age or older.

   3) Unresectable disease. Patients with resectable disease may be enrolled after having refused surgery after a documented consultation with a surgeon.

   4) Radiographic or visually measurable disease based on Response Evaluation Criteria In Solid Tumors, Version 1.1 criteria.

   5) At least one accessible primary or metastatic tumor site that can be readily injected IT with poly-ICLC with or without ultrasound guidance. This lesion can be superficial cutaneous, subcutaneous, or within a readily accessible location, including a lymph node, and must measure ≥ 15mm short axis for target.

   6) Patients who have received at least 8 weeks of aPD1 or aPDL1 immunotherapy and who have either progressive disease, stable disease or partial response based on RECIST 1.1 criteria are elegible for participation as separate cohorts B or C, with continuation of the aPD1 or aPDL1 therapy at their physician's discretion.

   7) ECOG performance status of ≤ 2. 8) Acceptable hematologic, renal and liver function as follows: A) Absolute neutrophil count > 1000/mm3 B) Platelets > 50,000/mm3, C) Creatinine ≤ 2.5 mg/dl, D) Total bilirubin ≤ 1.5 mg/dl, E) Transaminases ≤ 2 times above the upper limits of the institutional normal. F) INR<2 if off of anticoagulation. Patients on anticoagulation therapy with an INR>2 may be enrolled at the discretion of the investigator if they have not had any episodes of severe hemorrhage and if the site to be injected is not located in the oropharynx or another area where achieving homeostasis would be complicated by local anatomy.

   9) Patients must be able to provide informed consent. 10) Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception. Contraception must be continued for at least 2 months following the last dose of poly-ICLC. Women of childbearing potential must have a negative pregnancy test. While animal reproductive studies have been negative, the simulated viral infection and anti-proliferative activity of this experimental drug may theoretically affect the developing fetus or nursing infant.

   Cohort Specific Inclusion Criteria (see § 11.6 Evaluation of Best Overall Response (BOR)

   Cohort A) 11) Patients who are not receiving an anti-PD-1 or anti-PD-L1 agent,

   Cohort B 12) Patients who have received at least 8 weeks of aPD1 or aPDL1 immunotherapy. 13) Patients have progressive disease based on RECIST 1.1 criteria.

   Cohort C) 14) Patients who have received at least 8 weeks of aPD1 or aPDL1 immunotherapy. 15) Patients have stable disease or a partial response based on RECIST 1.1 criteria.

   4.2 Exclusion Criteria

   Patients with any of the following are ineligible for this research study:
   1. Serious concurrent infection or medical illness, which would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety.
   2. Bulky intracranial metastatic disease with shift of midline structures or progressive brain metastasis such that ongoing therapy for these brain metastasis is required at the time of enrollment.
   3. In the opinion of the local PI: Head and neck cancer patients with airway tumor recurrence that may compromise breathing or swallowing if inflammation or edema is transiently aggravated by Hiltonol® injection. Head and neck cancer patients with tumor invading major blood vessels for whom there may be a risk of blockage or bleeding if inflammation or edema is transiently increased by Hiltonol® injections.
   4. AIDS defined as a CD4 count less than 200 in the context of HIV sero-positivity or chronically is taking immunosuppressive medication such as steroids or transplant related medications.
   5. Life expectancy of less than 6 months in the judgment of the study physician.
   6. Persistent toxicity from recent therapy that has not sufficiently resolved in the judgment of the study physician.
   7. History of active cancer vaccine immunotherapy in the previous month. Patients who have received at least 8 weeks of aPD1 or aPDL1 immunotherapy and who have either progressive disease, stable disease or partial response based on RECIST 1.1 criteria are elegible for participation and continuation of the aPD1 or aPDL1 therapy at their physician's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-03; Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Evaluate safety of intratumoral (IT) plus intramuscular (IM) Polyinosinic-polycytidylic acid stabilized with polylysine and carboxymethylcellulose (poly-ICLC, Hiltonol®) for treatment of patients with accessible solid tumors, with or with | Evaluation of response wk 26
  Wk 26 study subject's response will be defined as BOR (CR, PR, SD) or PD.
Evaluate therapeutic efficacy assessed by Disease Control (CR, PR, or SD) as defined by the RECIST 1.1 Criteria. | 6 months
  Week 26 tumor assessment will be performed, an optional biopsy may be performed.

SECONDARY OUTCOMES:
Determine whether the study regimen of Poly-ICLC will induce an innate and/or an adaptive, specific anti-tumor T cell immune response in the injected tumor lesion and systemically. | 26 weeks
  Serial blood samples collected at certain time points and processed and used to evaluate humoral and cellular immunity induced by IT and IM polyICLC injections
Determine the response in injected lesions as defined by change in size at 16 weeks and 26 weeks as assessed by bi-dimensional measurement using RECIST 1.1 criteria. | 16 weeks and 26 weeks
  In the present protocol, we propose to induce both innate and adaptive cellular immune mechanisms with IT injections of poly-ICLC (Nierkens, den Brock et al. 2008)
Determine the response in non-injected tumor lesions, both visceral and non-visceral as defined by change in size at 16 weeks and 26 weeks as assessed by bi- dimensional measurement. | 16 weeks and 26 weeks
  Bi-dimensional measurements will be performed on injected and non-injected lesions at the indicated time points in the study calendar.
Determine progression free survival at 12, 24, and 36 months in treated study subjects. | 12, 24 and 36 months
  Up to 5 visible deep measureable lesions will be designated as Target Lesions (index lesions)
Determine overall survival (OS) in treated study subjects. | Up to 36 months
  Survival and disease control/progression-free survival (PFS) will be estimated using Kaplan-Meir curves.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Bhardwaj, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; David H Smith, MD, Principal Investigator — Bay Hematology Oncology; Kevin Staveley-O'Carroll, MD, Principal Investigator — University Missouri; Frederick P Smith, MD, Principal Investigator — Chevy Chase, RCCA
Locations (5):
- United States (5):
  - Chevy Chase RCCA, Chevy Chase, Maryland
  - Dermatologic Surgery Center Washington DC, Chevy Chase, Maryland
  - Bay Hematology Oncology, Easton, Maryland
  - University of Missouri School of Medicine, Columbia, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No
No plan to share data

REFERENCES:
- [Background] Bosio CM, Aman MJ, Grogan C, Hogan R, Ruthel G, Negley D, Mohamadzadeh M, Bavari S, Schmaljohn A. Ebola and Marburg viruses replicate in monocyte-derived dendritic cells without inducing the production of cytokines and full maturation. J Infect Dis. 2003 Dec 1;188(11):1630-8. doi: 10.1086/379199. Epub 2003 Nov 14. PMID 14639532
- [Background] Cella M, Salio M, Sakakibara Y, Langen H, Julkunen I, Lanzavecchia A. Maturation, activation, and protection of dendritic cells induced by double-stranded RNA. J Exp Med. 1999 Mar 1;189(5):821-9. doi: 10.1084/jem.189.5.821. PMID 10049946
- [Background] Cho HI, Celis E. Optimized peptide vaccines eliciting extensive CD8 T-cell responses with therapeutic antitumor effects. Cancer Res. 2009 Dec 1;69(23):9012-9. doi: 10.1158/0008-5472.CAN-09-2019. Epub 2009 Nov 10. PMID 19903852
- [Background] Davies ME, Field AK. Effect of poly I:C/poly-L-lysine (poly ICL) on the development of murine osteogenic sarcoma. J Interferon Res. 1983;3(1):89-95. doi: 10.1089/jir.1983.3.89. PMID 6573430
- [Background] Geiss G, Jin G, Guo J, Bumgarner R, Katze MG, Sen GC. A comprehensive view of regulation of gene expression by double-stranded RNA-mediated cell signaling. J Biol Chem. 2001 Aug 10;276(32):30178-82. doi: 10.1074/jbc.c100137200. PMID 11487589
- [Background] Houot R, Levy R. T-cell modulation combined with intratumoral CpG cures lymphoma in a mouse model without the need for chemotherapy. Blood. 2009 Apr 9;113(15):3546-52. doi: 10.1182/blood-2008-07-170274. Epub 2008 Oct 21. PMID 18941113
- [Background] Huang CC, Duffy KE, San Mateo LR, Amegadzie BY, Sarisky RT, Mbow ML. A pathway analysis of poly(I:C)-induced global gene expression change in human peripheral blood mononuclear cells. Physiol Genomics. 2006 Jul 12;26(2):125-33. doi: 10.1152/physiolgenomics.00002.2006. Epub 2006 Mar 22. PMID 16554548
- [Background] Kajiwara K, Morishima H, Akiyama K, Yanagihara Y. Expression and function of the inducible costimulator ligand B7-H2 in human airway smooth muscle cells. Allergol Int. 2009 Dec;58(4):573-83. doi: 10.2332/allergolint.09-OA-0113. Epub 2009 Sep 25. PMID 19776675
- [Background] Longhi MP, Trumpfheller C, Idoyaga J, Caskey M, Matos I, Kluger C, Salazar AM, Colonna M, Steinman RM. Dendritic cells require a systemic type I interferon response to mature and induce CD4+ Th1 immunity with poly IC as adjuvant. J Exp Med. 2009 Jul 6;206(7):1589-602. doi: 10.1084/jem.20090247. Epub 2009 Jun 29. PMID 19564349
- [Background] Marcus PI, Sekellick MJ. Combined sequential treatment with interferon and dsRNA abrogates virus resistance to interferon action. J Interferon Cytokine Res. 2001 Jun;21(6):423-9. doi: 10.1089/107999001750277907. PMID 11440640
- [Background] Morgan ET, Norman CA. Pretranslational suppression of cytochrome P-450h (IIC11) gene expression in rat liver after administration of interferon inducers. Drug Metab Dispos. 1990 Sep-Oct;18(5):649-53. PMID 1706245
- [Background] Nierkens S, den Brok MH, Sutmuller RP, Grauer OM, Bennink E, Morgan ME, Figdor CG, Ruers TJ, Adema GJ. In vivo colocalization of antigen and CpG [corrected] within dendritic cells is associated with the efficacy of cancer immunotherapy. Cancer Res. 2008 Jul 1;68(13):5390-6. doi: 10.1158/0008-5472.CAN-07-6023. PMID 18593941
- [Background] North RJ, Dunn PL, Havell EA. A role for tumor necrosis factor in poly(I:C)-induced hemorrhagic necrosis and T-cell-dependent regression of a murine sarcoma. J Interferon Res. 1991 Dec;11(6):333-40. doi: 10.1089/jir.1991.11.333. PMID 1839310
- [Background] Pilaro AM, Taub DD, McCormick KL, Williams HM, Sayers TJ, Fogler WE, Wiltrout RH. TNF-alpha is a principal cytokine involved in the recruitment of NK cells to liver parenchyma. J Immunol. 1994 Jul 1;153(1):333-42. PMID 8207246
- [Background] Salazar AM, Levy HB, Ondra S, Kende M, Scherokman B, Brown D, Mena H, Martin N, Schwab K, Donovan D, Dougherty D, Pulliam M, Ippolito M, Graves M, Brown H, Ommaya A. Long-term treatment of malignant gliomas with intramuscularly administered polyinosinic-polycytidylic acid stabilized with polylysine and carboxymethylcellulose: an open pilot study. Neurosurgery. 1996 Jun;38(6):1096-103; discussion 1103-4. PMID 8727138
- [Background] Salem ML, El-Naggar SA, Kadima A, Gillanders WE, Cole DJ. The adjuvant effects of the toll-like receptor 3 ligand polyinosinic-cytidylic acid poly (I:C) on antigen-specific CD8+ T cell responses are partially dependent on NK cells with the induction of a beneficial cytokine milieu. Vaccine. 2006 Jun 12;24(24):5119-32. doi: 10.1016/j.vaccine.2006.04.010. Epub 2006 May 2. PMID 16704888
- [Background] Sivori S, Falco M, Della Chiesa M, Carlomagno S, Vitale M, Moretta L, Moretta A. CpG and double-stranded RNA trigger human NK cells by Toll-like receptors: induction of cytokine release and cytotoxicity against tumors and dendritic cells. Proc Natl Acad Sci U S A. 2004 Jul 6;101(27):10116-21. doi: 10.1073/pnas.0403744101. Epub 2004 Jun 24. PMID 15218108
- [Background] Stahl-Hennig C, Eisenblatter M, Jasny E, Rzehak T, Tenner-Racz K, Trumpfheller C, Salazar AM, Uberla K, Nieto K, Kleinschmidt J, Schulte R, Gissmann L, Muller M, Sacher A, Racz P, Steinman RM, Uguccioni M, Ignatius R. Synthetic double-stranded RNAs are adjuvants for the induction of T helper 1 and humoral immune responses to human papillomavirus in rhesus macaques. PLoS Pathog. 2009 Apr;5(4):e1000373. doi: 10.1371/journal.ppat.1000373. Epub 2009 Apr 10. PMID 19360120
- [Background] van der Most RG, Currie A, Robinson BW, Lake RA. Cranking the immunologic engine with chemotherapy: using context to drive tumor antigen cross-presentation towards useful antitumor immunity. Cancer Res. 2006 Jan 15;66(2):601-4. doi: 10.1158/0008-5472.CAN-05-2967. PMID 16423984
- [Background] Wong JP, Christopher ME, Viswanathan S, Dai X, Salazar AM, Sun LQ, Wang M. Antiviral role of toll-like receptor-3 agonists against seasonal and avian influenza viruses. Curr Pharm Des. 2009;15(11):1269-74. doi: 10.2174/138161209787846775. PMID 19355966
- [Background] Zhu X, Nishimura F, Sasaki K, Fujita M, Dusak JE, Eguchi J, Fellows-Mayle W, Storkus WJ, Walker PR, Salazar AM, Okada H. Toll like receptor-3 ligand poly-ICLC promotes the efficacy of peripheral vaccinations with tumor antigen-derived peptide epitopes in murine CNS tumor models. J Transl Med. 2007 Feb 12;5:10. doi: 10.1186/1479-5876-5-10. PMID 17295916
- [Derived] Kyi C, Roudko V, Sabado R, Saenger Y, Loging W, Mandeli J, Thin TH, Lehrer D, Donovan M, Posner M, Misiukiewicz K, Greenbaum B, Salazar A, Friedlander P, Bhardwaj N. Therapeutic Immune Modulation against Solid Cancers with Intratumoral Poly-ICLC: A Pilot Trial. Clin Cancer Res. 2018 Oct 15;24(20):4937-4948. doi: 10.1158/1078-0432.CCR-17-1866. Epub 2018 Jun 27. PMID 29950349